CLINICAL TRIAL: NCT05679687
Title: A Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of Allogeneic Anti CD19 CAR-T Bridging to Hematopoietic Stem Cell Transplantation in Patients With Refractory or Relapsed B Cell Acute Lymphoblastic Leukemia
Brief Title: ThisCART19A Bridging to alloHSCT for R/R B-ALL
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: Fundamenta Therapeutics, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SZ4602
Record Dates: First submitted 2022-12-27; First posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-12

CONDITIONS: CAR; Refractory Acute Lymphoblastic Leukemia; Relapsed Adult ALL
Keywords: Universal CAR-T; allogeneic HCT
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): In this study, allogeneic anti-CD19 CAR T cells (ThisCART19A) infusion is used as a bridge therapy to hematopoietic stem cell transplantation to treat patients with refractory or relapsed CD19 positive B cell acute lymphoblastic leukemia. Lymphodepletion conditioning before CAR T cell infusion consists of fludarabine, CTX and VP-16.
  Interventions: Drug: Treatment

INTERVENTIONS:
Drug: Treatment — In this study, allogeneic anti-CD19 CAR T cells (ThisCART19A) infusion is used as a bridge therapy to hematopoietic stem cell transplantation to treat patients with refractory or relapsed CD19 positive B cell acute lymphoblastic leukemia. Lymphodepletion conditioning before CAR T cell infusion consists of fludarabine, CTX and VP-16.

SUMMARY:
This is a phase 1, open-label study to assess the efficacy, safety and pharmacokinetics of ThisCART19A (Allogeneic Anti CD19 CAR-T) bridging to HSCT in patients with refractory or relapsed B cell acute lymphoblastic leukemia (r/r B-ALL).

DETAILED DESCRIPTION:
This is a phase 1, single-center, nonrandomized, open-label, dose-escalation study to evaluate the efficacy, safety and pharmacokinetics of ThisCART19A bridging to HSCT in patients with CD19 positive r/r B-ALL and identify a treatment regimen most likely to result in clinical efficacy while maintaining a favorable safety profile. Before initiating ThisCART19A infusion, subjects will be administered lymphodepletion chemotherapy composed of fludarabine、cyclophosphamide and VP-16. At Day 0 of the Treatment Period, subjects will receive an intravenous (IV) infusion of ThisCART19A. All subjects are monitored during the treatment period through Day 28. All subjects who receive a dose of ThisCART19A will be followed up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign a documented IRB-approved ICF prior to any screening procedure.
2. No gender limitation, 14 years ≤ age ≤ 65 years.
3. Intention to HSCT therapy.
4. Meeting the diagnostic criteria of relapsed or refractory B-ALL. Relapsed B-ALL: Reappearance of blasts in the blood or bone marrow (>5%) or in any extramedullary site after a CR. Refractory B-ALL: Failure to achieve CR or CRi at the end of induction therapy (General refers to a 4-week regimen or a Hyper-CVAD regimen); Subjects with Ph+ disease are eligible if they are intolerant to TKI therapy, or if they have relapsed/refractory disease despite treatment with at least 2 different TKIs.
5. Life expectancy ≥ 8 weeks at the time of enrollment.
6. Eastern Cooperative Oncology Group performance status score of 0 or 1.
7. Adequate bone marrow, renal, hepatic, pulmonary and cardiac function:

   1. Adequate marrow function for lymphodepletion chemotherapy assessed by the investigator.
   2. Creatinine clearance > 30 mL/min according to the Cockcroft-Gault formula;
   3. ALT and AST ≤ 5 × ULN (the upper limit of normal), total bilirubin ≤ 2×ULN. (Subjects with Gilbert syndrome or liver involvement may be included if their total bilirubin is ≤ 3 × ULN.)
   4. Oxygen saturation (SaO2) ≥ 92% on room air.
   5. Cardiac function：left ventricular ejection fraction (LVEF) ≥ 40% assessed by echocardiography.
8. CD19-positive leukemia obtained from bone marrow or peripheral blood confirmed by flowcytometry or biopsy during screening.

Exclusion Criteria:

1. Allergic to preconditioning measures.
2. History of allogeneic HSCT.
3. Other malignancies apart from B-cell malignancies within 5 years prior to screening. (Subjects with cured skin squamous carcinoma, basal cell carcinoma, non-primary invasive bladder cancer, localized low-risk prostate cancer, in situ cervical/breast cancer can be enrolled.)
4. Severe active infection. (Simple urinary tract infection (UTI) and uncomplicated bacterial pharyngitis are permitted.)
5. Pulmonary embolism within 3 months prior to enrollment.
6. Severe cardiovascular and cerebrovascular diseases and hereditary diseases intolerant to CAR-T therapy assessed by the investigator prior to enrollment.
7. Presence of symptomatic CNS involvement (both primary and secondary) at screening confirmed by imaging;
8. Active hepatitis B virus (defined as serum HBV-DNA ≥ 2000 IU/mL), hepatitis C virus (HCV), human immunodeficiency virus (HIV) or active syphilis infection prior to enrollment. (Subjects with HBV-DNA < 2000 IU/mL can be enrolled, but should be administered antiviral drugs such as entecavir and tenofovir with relative clinical indicators monitored simultaneously during the treatment.)
9. Vaccinated with influenza vaccine within 2 weeks prior to lymphodepletion chemotherapy. (Subjects vaccinated with SARS-COV19 vaccine or inactivated, live/non-live adjuvant vaccines can be enrolled.)
10. Female subjects who are pregnant, breastfeeding or planning for pregnancy within 1 year after CAR-T cell infusion, or male subjects whose partners are planning for pregnancy within 1 year after CAR-T cell infusion.
11. Any conditions that would, in the investigator's assessment, increase risks in patients or interfere with the outcomes of the trial.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
ORR | 4 week
  Overall response rate
MRD Negativity | 4 week
  MRD Negativity is assessed utilizing multicolor flow cytometry to detect leukemia cells with a sensitivity of 10^ (-4).

SECONDARY OUTCOMES:
CR | 2 year
  Complete response
CRi | 2 year
  CR with incomplete hematologic recovery
CRh | 2 year
  CR with partial hematological recovery
BFBM | 2 year
  Blast-free hypoplastic or aplastic bone marrow
PR | 2 year
  Partial response
DOR | 2 year
  Duration of response
LFS | 2 year
  Leukemia-free survival
OS | 2 year
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided